CLINICAL TRIAL: NCT01903031
Title: Evaluating Pharmacokinetic Interactions With Vaginal Ring Contraceptives and Antiretroviral Therapy (ART)
Brief Title: Evaluating Pharmacokinetic Interactions With Vaginal Ring Contraceptives and ART
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5316; UM1AI068636 (NIH)
Record Dates: First submitted 2013-07-16; First posted 2013-07-19 (Estimated); Results first posted 2018-01-04 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — efavirenz; atazanavir, ritonavir drug combination; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- NuvaRing and no ART (Arm A) (Experimental): Once NuvaRing is inserted into the vagina, the ring should remain in place (not be removed) continuously for 3 weeks (21 days).
  Interventions: Device: Nuvaring
- NuvaRing with EFV plus ≥2 NRTIs (Arm B) (Experimental): Once NuvaRing is inserted into the vagina, the ring should remain in place (not be removed) continuously for 3 weeks (21 days). EFV is a non-nucleoside reverse transcriptase inhibitor taken at a dose of 600 mg once daily.
  Interventions: Device: Nuvaring; Drug: EFV; Drug: NRTIs
- NuvaRing with ATV/r plus TDF + ≥1 NRTIs (Arm C) (Experimental): Once NuvaRing is inserted into the vagina, the ring should remain in place (not be removed) continuously for 3 weeks (21 days). ATV/r is a combination protease inhibitor taken at a dose of 300/100 mg once daily. Tenofovir disoproxil fumarate (TDF) is a nucleoside reverse transcriptase inhibitor (NRTI) taken at a dose of 300 mg daily.
  Interventions: Device: Nuvaring; Drug: ATV/r; Drug: TDF; Drug: NRTIs

INTERVENTIONS:
Device: Nuvaring — NuvaRing is made of ethylene vinylacetate copolymers (28% and 9% vinylacetate) and magnesium stearate, is latex free, and contains 11.7 mg etonogestrel and 2.7 mg ethinyl estradiol. NuvaRing has an outer diameter of 54 mm and a cross-sectional diameter of 4mm. Once NuvaRing is inserted into the vagina, the ring should remain in place (not be removed) continuously for 3 weeks (21 days). After being in place for the first 21 days of the study, the ring may be removed after the day 21 study visit evaluations have been completed.
  Other Names: Etonogestrel/ethinyl estradiol vaginal ring
Drug: EFV — Participants received EFV 600 mg daily with two or more NRTIs
  Other Names: Efavirenz
  Arms: NuvaRing with EFV plus ≥2 NRTIs (Arm B)
Drug: ATV/r — Participants received ATV/r 300 mg/ 100 mg daily with tenofovir and one or more additional NRTIs
  Other Names: Atazanavir/Ritonavir
  Arms: NuvaRing with ATV/r plus TDF + ≥1 NRTIs (Arm C)
Drug: TDF — Participants received 300 mg of tenofovir in Arm C
  Other Names: Tenofovir Disoproxil Fumarate
  Arms: NuvaRing with ATV/r plus TDF + ≥1 NRTIs (Arm C)
Drug: NRTIs — Participants received two or more NRTIs in Arm B and one or more NRTIs in Arm C
  Other Names: Nucleoside Reverse Transcriptase Inhibitor
  Arms: NuvaRing with ATV/r plus TDF + ≥1 NRTIs (Arm C); NuvaRing with EFV plus ≥2 NRTIs (Arm B)

SUMMARY:
This study was done to look at a method of hormonal birth control, called the NuvaRing, and specific anti-HIV medications, called antiretrovirals (ARVs). Some studies of women who use a hormonal birth control method (specifically oral pills, patches, and injections) and take ARVs have shown that ARVs interact with the hormones released by the birth control medication. These interactions may cause the birth control to be less effective at preventing pregnancy. There is also concern that hormonal birth control can increase HIV spreading to others, but more studies are needed to determine if this is true. The investigators did not know whether the NuvaRing and ARVs interact when they are used together, so this study looked to see if certain ARVs (efavirenz and atazanavir/ritonavir) interact with the two hormones released by NuvaRing. This will help us to determine if NuvaRing is safe and effective for women with HIV infection who are taking ARVs. The study also included HIV-infected women who were not on ARVs but used the NuvaRing to show us what the hormone levels are like in a similar group of women not on ARVs.

Vaginal rings are also currently being studied to deliver anti-HIV medications that may prevent HIV acquisition, and to provide birth control over a longer period of time (more than 1 month). Since vaginal rings will become more commonly used to administer medications, the investigators wanted to better understand the potential for drug interactions with drugs given vaginally. This study will also help us understand the potential for drug interactions between ARVs given orally, and other drugs given through vaginal rings, like the NuvaRing. Additionally, this study will help us understand how hormones released from a vaginal ring affect the amount of HIV virus in the genital tract, the bacterial make-up (microbiome) of the female genital tract, and the immune system within the genital tract, all of which may affect the chances of spreading HIV.

DETAILED DESCRIPTION:
This was a 28 day study from study entry through the final clinic visit. Post-entry visits were scheduled at Days 7, 14, 21 and 28. The Nuvaring was put in place at study entry and removed on day 21. A single pharmacokinetic (PK) blood sample was collected for assay of etonogestrel (ENG) and ethinyl estradiol (EE) at entry (day 0, prior to NuvaRing placement), and on days 7, 14, and 21 after placement of the NuvaRing. For participants on the ARV arms, intensive, 8-hour PK sampling, for assay of efavirenz (EFV) and atazanavir/ritonavir (ATV/RTV) respectively, was performed at study entry (day 0, prior to NuvaRing placement) and 21 days later. ARV sampling was performed at pre-dose (hour 0), and 1, 3, 4, 5, and 8 hours post-dose. Safety was assessed at each study visit.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection.
* Participants must have been receiving either 1) EFV 600 mg daily with 2 or more NRTIs, 2) ATV/r 300 mg/ 100 mg daily with TDF 300 mg and 1 or more additional NRTIs, or 3) no ART. ART regimens should have been stable for 30 days prior to study entry with no plans to change therapy during the first 28 days of this study. Participants receiving no ART should have had no plans to initiate ART during the first 28 days of the study.

NOTE: Participants must have had access to their ART regimens through their primary care providers. ART medications were not supplied by this study.

* For participants on ART, documentation of plasma HIV-1 RNA ≤400 copies/mL was obtained within 60 days prior to study entry.
* For participants not on ART, CD4+ cell count must have been ≥350 cells/mm^3, obtained within 60 days prior to study entry.
* Laboratory values within 60 days prior to study entry:

  * Platelet count ≥50,000 platelets/mm^3
  * Hemoglobin ≥8.0 g/dL
  * Aspartate transaminase (SGOT) and alanine aminotransferase (SGPT) <5 x upper limit of normal (ULN)
  * Creatinine ≤1.5 x ULN
  * Total bilirubin ≤2.0 x ULN
* Last menstrual period ≤6 months prior to study entry. If last menstrual period >6 months prior to study entry without another cause for amenorrhea, such as recent pregnancy, serum follicle-stimulating hormone (FSH) must have been checked and be ≤40 mIU/mL to be eligible for enrollment.
* Premenopausal females with at least one functioning ovary.
* Documentation of Pap smear within 1 year prior to study entry.
* Negative serum or urine-HCG pregnancy test with a sensitivity of ≤25 mIU/mL within 60 days prior to study entry and within 24 hours prior to study entry
* All participants must have agreed not to participate in a conception process (eg, active attempt to become pregnant or in vitro fertilization) for the duration of the study. Because it was unknown if ARVs adversely affect the efficacy of NuvaRing as a contraceptive method, participants of reproductive potential, who were participating in sexual activities that could lead to pregnancy, must have agreed to use an additional reliable form of contraception while in the study. Acceptable additional methods of contraception included:

  * Condoms (male or female)
  * Non-hormonal intrauterine device (IUD)

Other hormonal forms of contraception were not allowed during the study period.

Condoms should have been used to prevent transmission of HIV and sexually transmitted diseases between sexual partners.

NOTE: Participants with bilateral tubal ligation or non-hormonal IUD were eligible to be enrolled.

Exclusion Criteria:

* Received depot medroxyprogesterone acetate (DMPA) within 4 months prior to study entry.
* Received other hormonal therapies (eg, oral contraceptive agents, hormone- containing vaginal ring, contraceptive patch, hormone replacement therapy, anabolic therapies, including nandrolone decanoate or megestrol acetate) within 30 days prior to study entry.
* Breastfeeding.
* Less than 6 weeks postpartum at study entry.
* Use of any prohibited medications within 30 days prior to study entry.
* Initiated, discontinued, or changed doses of drugs that are CYP substrates or known to have drug interactions with ethinyl estradiol or etonogestrel within 30 days prior to study entry.
* Bilateral oophorectomy.
* For women older than 35 years of age, smoking 15 or more cigarettes per day.
* History of invasive cancer of the reproductive tract; known or suspected malignancy of the breast, or known increased risk for breast cancer; undiagnosed abnormal vaginal bleeding; liver tumors; or serious ocular disorders at any time prior to study entry.
* Chronic immunosuppressive conditions other than HIV.
* Use of systemic or inhaled corticosteroids such as for acute therapy for Pneumocystis pneumonia (PCP) or asthma exacerbation and prednisone ≥10 mg (or equivalent) for any reason other than a stable or tapering dose.
* History of deep venous thrombosis or pulmonary embolism.
* History of cerebral vascular or coronary artery disease.
* Severe uncontrolled hypertension within 60 days prior to study entry.
* Diabetes with vascular involvement.
* Clinically active cervical or vaginal infection at study entry. NOTE: Gonorrhea, chlamydia, and trichomonas testing was performed during screening using techniques available at the local sites and documented in source documentation and case report forms (CRFs). Testing for bacterial vaginosis, performed using techniques available at the local sites, was only necessary if the participant was symptomatic and the provider felt treatment might be necessary. Women with genital herpes lesions waited to be screened until the herpetic lesions had healed.
* Acute infections or other opportunistic diseases requiring medication within 14 days prior to study entry.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2014-12-30 (Actual); Primary Completion 2016-10-03 (Actual); Study Completion 2016-10-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (10):
  - 31788 Alabama CRS, Birmingham, Alabama
  - University of Southern California LA (5048), Los Angeles, California
  - David Geffen School of Medicine at UCLA NICHD CRS (5112), Los Angeles, California
  - University of Colorado Denver NICHD CRS (5052), Aurora, Colorado
  - University of Florida Jacksonville (5051), Jacksonville, Florida
  - Rush University Cook County Hospital Chicago NICHD CRS (5083), Chicago, Illinois
  - 31786 New Jersey Medical School Clinical Research Center CRS, Newark, New Jersey
  - Columbia Physicians and Surgeons CRS (30329), New York, New York
  - Jacobi Medical Center Bronx, The Bronx, New York
  - The Miriam Hosp. ACTG CRS (2951), Providence, Rhode Island
- Gaborone Prevention/Treatment Trials CRS (12701), Gaborone, Botswana
- Instituto de Pesquisa Clinica Evandro Chagas (12101), Rio de Janeiro, Brazil
- Kenya Medical Research Institute/Center for Disease Control (KEMRI/CDC) CRS (31460), Kisumu, Kenya
- Peru (2):
  - Investigaciones Medicas en Salud (INMENSA) (11302), San Isidro, Lima region
  - Asociacion Civil Impacta Salud y Educacion - Miraf CRS (11301), Lima
- Puerto Rico (3):
  - Puerto Rico-AIDS CRS (5401), San Juan
  - University of Puerto Rico Pediatric HIV/AIDS Research Program CRS (6601), San Juan
  - San Juan Hospital PR NICHD CRS (5031), San Juan
- Shandukani Research CRS (8051), Johannesburg, Gauteng, South Africa
- Thailand (2):
  - 31802 Thai Red Cross AIDS Research Center Treatment (TRC-ARC Treatment) CRS, Bangkok, Patumwan
  - 31784 Chiang Mai University HIV Treatment CRS, Chiang Mai

REFERENCES:
- [Derived] Scarsi KK, Cramer YS, Rosenkranz SL, Aweeka F, Berzins B, Coombs RW, Coughlin K, Moran LE, Zorrilla CD, Akelo V, Aziz M, Friedman RK, Gingrich D, Swaminathan S, Godfrey C, Cohn SE; AIDS Clinical Trials Group A5316 Study Team. Antiretroviral therapy and vaginally administered contraceptive hormones: a three-arm, pharmacokinetic study. Lancet HIV. 2019 Sep;6(9):e601-e612. doi: 10.1016/S2352-3018(19)30155-9. PMID 31498109
- See also: Location of DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004 (Clarification, August 2009). — http://rsc.tech-res.com/safetyandpharmacovigilance/
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — http://rsc.tech-res.com/clinical-research-sites/safety-reporting/manual

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant enrolled in December 2014 and final participant enrolled in September 2016. Enrollment took place at 21 US and non-US clinical research sites.
Groups:
- NuvaRing and no ART: Participants who were not on ART were prescribed NuvaRing, to be inserted at entry and removed at Day 21.
- NuvaRing With EFV Plus ≥2 NRTIs: NuvaRing was inserted at entry and removed at Day 21. Participants also received EFV 600 mg daily with two or more NRTIs.
- NuvaRing With ATV/r Plus TDF and ≥1 NRTIs: NuvaRing was inserted at entry and removed at Day 21. Participants also received ATV/r 300 mg/ 100 mg daily with tenofovir (TDF) 300 mg and 1 or more additional NRTIs.
Period: Overall Study
Arm/Group | NuvaRing and no ART | NuvaRing With EFV Plus ≥2 NRTIs | NuvaRing With ATV/r Plus TDF and ≥1 NRTIs
Started | 27 | 28 | 29
Completed | 25 | 25 | 24
Not Completed | 2 | 3 | 5
Not completed — Not Able to Attend Clinic | 1 | 1 | 0
Not completed — Missed Day 21 Primary Endpoint Visit | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — NuvaRing removed prior to Day 21 visit | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | NuvaRing and no ART | NuvaRing With EFV Plus ≥2 NRTIs | NuvaRing With ATV/r Plus TDF and ≥1 NRTIs | Total
Number analyzed (Participants) | 27 | 28 | 29 | 84
Age, Continuous [Median (Full Range); unit: years] | 32 [22 to 48] | 36 [17 to 55] | 36 [22 to 50] | 35 [17 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 28 | 29 | 84
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 1 | 1 | 1 | 3
  Black Non-Hispanic | 12 | 18 | 14 | 44
  Hispanic (Regardless of Race) | 11 | 9 | 9 | 29
  Asian, Pacific Islander | 3 | 0 | 5 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  Puerto Rico | 1 | 0 | 2 | 3
  United States | 5 | 14 | 15 | 34
  Botswana | 4 | 1 | 0 | 5
  Brazil | 3 | 6 | 5 | 14
  South Africa | 2 | 0 | 0 | 2
  Kenya | 3 | 3 | 2 | 8
  Thailand | 3 | 0 | 5 | 8
  Peru | 6 | 4 | 0 | 10

OUTCOME MEASURES:

1. Primary Outcome: Etonogestrel Concentrations at Study Day 21
Description: This evaluates the effect of EFV and ATV/r on etonogestrel by measuring etonogestrel concentrations on all three study arms 21 days after NuvaRing administration. The pharmacokinetic (PK) blood sample for measurement of etonogestrel on study day 21 was taken before the NuvaRing was removed. The assay lower limit of quantification for etonogestrel was 250 pg/mL; values < 250 were assigned a value of half the lower limit (ie, 125 pg/mL).
Time Frame: Day 21
Population: Participants who provided the Etonogestrel PK sample at day 21 were included in the analysis.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | NuvaRing and no ART | NuvaRing With EFV Plus ≥2 NRTIs | NuvaRing With ATV/r Plus TDF and ≥1 NRTIs
Number analyzed (Participants) | 25 | 25 | 24
pg/mL | 1860.00 [665.00 to 3590.00] | 429.00 [125.00 to 1180.00] | 3290.00 [730.00 to 6920.00]
Statistical Analysis 1: Comparison: NuvaRing and no ART vs NuvaRing With EFV Plus ≥2 NRTIs; Null hypothesis: There is no difference in concentrations of Etonogestrel on day 21 between the control arm (NuvaRing and no ART) and NuvaRing with EFV plus ≥2 NRTIs; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons were made. Statistical significance was declared if p<0.05
Statistical Analysis 2: Comparison: NuvaRing and no ART vs NuvaRing With ATV/r Plus TDF and ≥1 NRTIs; Null hypothesis: There is no difference in concentrations of Etonogestrel on day 21 between the control arm (NuvaRing and no ART) and NuvaRing with ATV/r plus TDF and ≥1 NRTIs; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons were made. Statistical significance was declared if p<0.05

2. Primary Outcome: Ethinyl Estradiol Concentrations at Study Day 21
Description: This evaluates the effect of EFV and ATV/r on ethinyl estradiol by measuring ethinyl estradiol concentrations on all three study arms 21 days after NuvaRing administration. The PK blood sample for measurement of ethinyl estradiol on study day 21 was taken before the NuvaRing was removed. The assay lower limit of quantification for ethinyl estradiol was 5 pg/mL ; values < 5 were assigned a value of half the lower limit (ie, 2.5 pg/mL).
Time Frame: Day 21
Population: Participants who provided the Ethinyl Estradiol PK sample at day 21 were included in the analysis.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | NuvaRing and no ART | NuvaRing With EFV Plus ≥2 NRTIs | NuvaRing With ATV/r Plus TDF and ≥1 NRTIs
Number analyzed (Participants) | 25 | 25 | 24
pg/mL | 21.30 [6.46 to 51.00] | 11.40 [2.50 to 21.00] | 16.05 [2.50 to 26.40]
Statistical Analysis 1: Comparison: NuvaRing and no ART vs NuvaRing With EFV Plus ≥2 NRTIs; Null hypothesis: There is no difference in concentrations of Ethinyl Estradiol on day 21 between the control arm (NuvaRing and no ART) and NuvaRing with EFV plus ≥2 NRTIs; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons were made. Statistical significance was declared if p<0.05
Statistical Analysis 2: Comparison: NuvaRing and no ART vs NuvaRing With ATV/r Plus TDF and ≥1 NRTIs; Null hypothesis: There is no difference in concentrations of Ethinyl Estradiol on day 21 between the control arm (NuvaRing and no ART) and NuvaRing with ATV/r plus TDF and ≥1 NRTIs; Test type: Other; p = 0.004, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons were made. Statistical significance was declared if p<0.05

3. Secondary Outcome: Etonogestrel Concentrations Obtained on Study Days 7 and 14
Description: This evaluates the effect of EFV and ATV/r on etonogestrel by measuring etonogestrel concentrations on all three study arms 7 and 14 days after NuvaRing administration. The assay lower limit of quantification for etonogestrel was 250 pg/mL; values < 250 were assigned a value of half the lower limit (ie, 125 pg/mL).
Time Frame: Study days 7 and 14
Population: Participants who provided the Etonogestrel PK samples at day 7 and at day 14 were included in the analysis.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | NuvaRing and no ART | NuvaRing With EFV Plus ≥2 NRTIs | NuvaRing With ATV/r Plus TDF and ≥1 NRTIs
Number analyzed (Participants) | 25 | 25 | 24
pg/mL
  Concentration at Day 7: number analyzed (Participants) | 24 | 25 | 24
  Concentration at Day 7 | 1970.00 [703.00 to 3220.00] | 427.00 [125.00 to 916.00] | 3250.00 [1330.00 to 4960.00]
  Concentration at Day 14: number analyzed (Participants) | 23 | 25 | 24
  Concentration at Day 14 | 2070.00 [648.00 to 3720.00] | 437.00 [125.00 to 1090.00] | 3530.00 [725.00 to 6100.00]

4. Secondary Outcome: Ethinyl Estradiol Concentrations Obtained on Study Days 7 and 14.
Description: This evaluates the effect of EFV and ATV/r on ethinyl estradiol by measuring ethinyl estradiol concentrations on all three study arms 7 and 14 days after NuvaRing administration. The assay lower limit of quantification for ethinyl estradiol was 5 pg/mL; values < 5 were assigned a value of half the lower limit (ie, 2.5 pg/mL).
Time Frame: Study days 7 and 14
Population: Participants who provided the Ethinyl estradiol PK samples at day 7 and at day 14 were included in the analysis.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | NuvaRing and no ART | NuvaRing With EFV Plus ≥2 NRTIs | NuvaRing With ATV/r Plus TDF and ≥1 NRTIs
Number analyzed (Participants) | 25 | 25 | 24
pg/mL
  Concentration at Day 7: number analyzed (Participants) | 24 | 25 | 24
  Concentration at Day 7 | 18.05 [6.71 to 50.90] | 9.98 [2.50 to 18.70] | 15.70 [5.48 to 24.30]
  Concentration at Day 14: number analyzed (Participants) | 23 | 25 | 24
  Concentration at Day 14 | 19.70 [6.51 to 47.90] | 10.50 [2.50 to 18.60] | 16.55 [6.76 to 26.90]

5. Secondary Outcome: EFV PK Parameter Area Under the Concentration-Time Curve (AUC0-24hours) Calculated Based on Intensive EFV PK Samples Obtained From Individual Participants Enrolled in Arm B
Description: This evaluates the effect of NuvaRing on the PK parameter AUC(0-24h) of EFV before NuvaRing placement (at study day 0) and three weeks later (on study day 21), prior to NuvaRing removal. AUC(0-24h) defines area under the concentration-time curve over the period of 24 hours (pre-dose concentration was used to impute concentration at 24h).
Time Frame: Intensive EFV PK samples at pre-dose, 1, 3, 4, 5, and 8 hours post-dose on study day 0 (before vaginal ring placement) and on study day 21 (3 weeks after vaginal ring placement).
Population: The analysis population is the 24 A5316 participants enrolled in Arm B (NuvaRing with EFV arm plus 2 or more NRTIs) eligible for the secondary outcome of EFV PK parameters.
Measure: Median (Full Range); unit: h*ng/mL
Arm/Group | NuvaRing With EFV Plus ≥2 NRTIs
Number analyzed (Participants) | 24
h*ng/mL
  AUC0-24h day 0 | 68949.1 [27114.3 to 367995.4]
  AUC0-24h day 21 | 57795.9 [26326.3 to 362821.3]

6. Secondary Outcome: EFV PK Parameter Minimum Plasma Concentration (Cmin) Determined Based on EFV Levels From Individual Participants Enrolled in Arm B
Description: This evaluates the effect of NuvaRing on the EFV PK parameter Cmin obtained from both sampling periods, before NuvaRing placement (at study day 0) and three weeks later (on study day 21), prior to NuvaRing removal. Cmin defines minimum concentration observed within the first 8 hours of the 24 hour dosing interval.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Median (Full Range); unit: ng/mL
Arm/Group | NuvaRing With EFV Plus ≥2 NRTIs
Number analyzed (Participants) | 24
ng/mL
  Cmin day 0 | 2121.5 [903.7 to 13620.0]
  Cmin day 21 | 1766.0 [10.0 to 12930.0]

7. Secondary Outcome: EFV PK Parameter Maximum Plasma Concentration (Cmax) Determined Based on EFV Levels From Individual Participants Enrolled in Arm B
Description: This evaluates the effect of NuvaRing on the EFV PK parameter Cmax obtained from both sampling periods, before NuvaRing placement (at study day 0) and three weeks later (on study day 21), prior to NuvaRing removal. Cmax defines maximum concentration observed within the first 8 hours of the 24 hour dosing interval.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Median (Full Range); unit: ng/mL
Arm/Group | NuvaRing With EFV Plus ≥2 NRTIs
Number analyzed (Participants) | 24
ng/mL
  Cmax day 0 | 4541.0 [1347.0 to 18670.0]
  Cmax day 21 | 3786.0 [2231.0 to 19110.0]

8. Secondary Outcome: EFV PK Parameter Clearance (CLss/F) Determined Based on EFV Levels From Individual Participants Enrolled in Arm B
Description: This evaluates the effect of NuvaRing on the EFV PK parameter CLss/F obtained from both sampling periods, before NuvaRing placement (at study day 0) and three weeks later (on study day 21), prior to NuvaRing removal. CLss/F defines apparent oral clearance
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Median (Full Range); unit: L/h
Arm/Group | NuvaRing With EFV Plus ≥2 NRTIs
Number analyzed (Participants) | 24
L/h
  CLss/F day 0 | 8.7 [1.6 to 22.1]
  CLss/F day 21 | 10.4 [1.7 to 22.8]

9. Secondary Outcome: ATV PK Parameter AUC(0-24h) Calculated Based on Intensive Atazanavir (ATV) PK Samples Obtained From Individual Participants Enrolled in Arm C
Description: This evaluates the effect of NuvaRing on the PK parameter AUC(0-24h) of ATV before NuvaRing placement (at study day 0) and three weeks later (on study day 21), prior to NuvaRing removal. AUC(0-24h) defines area under the concentration-time curve over the period of 24 hours (pre-dose concentration was used to impute concentration at 24h).
Time Frame: Intensive ATV PK samples at pre-dose, 1, 3, 4, 5, and 8 hours post-dose on study day 0 (before vaginal ring placement) and on study day 21 (3 weeks after vaginal ring placement)
Population: The analysis population is the 23 A5316 participants enrolled in Arm C (NuvaRing with ATV/r arm plus TDF and one or more NRTIs) eligible for the secondary outcome of ATV PK parameters.
Measure: Median (Full Range); unit: h*ng/mL
Arm/Group | NuvaRing With ATV/r Plus TDF and ≥1 NRTIs
Number analyzed (Participants) | 23
h*ng/mL
  AUC0-24h day 0 | 44313.7 [8802.3 to 91766.5]
  AUC0-24h day 21 | 36764.7 [1346.9 to 108450.6]

10. Secondary Outcome: ATV PK Parameter Cmin Determined Based on ATV Levels From Individual Participants Enrolled in Arm C
Description: This evaluates the effect of NuvaRing on the ATV PK parameter Cmin obtained from both sampling periods, before NuvaRing placement (at study day 0) and three weeks later (on study day 21), prior to NuvaRing removal. Cmin defines minimum concentration observed within the first 8 hours of the 24 hour dosing interval.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Median (Full Range); unit: ng/mL
Groups:
- NuvaRing With ATV/r Plus TDF ≥1 NRTIs: NuvaRing was inserted at entry and removed at Day 21. Participants also received ATV/r 300 mg/ 100 mg daily with tenofovir (TDF) 300 mg and 1 or more additional NRTIs.
Arm/Group | NuvaRing With ATV/r Plus TDF ≥1 NRTIs
Number analyzed (Participants) | 23
ng/mL
  Cmin day 0 | 796.7 [10.0 to 2731.0]
  Cmin day 21 | 599.4 [10.0 to 3599.0]

11. Secondary Outcome: ATV PK Parameter Cmax Determined Based on ATV Levels From Individual Participants Enrolled in Arm C
Description: This evaluates the effect of NuvaRing on the ATV PK parameter Cmax obtained from both sampling periods, before NuvaRing placement (at study day 0) and three weeks later (on study day 21), prior to NuvaRing removal. Cmax defines maximum concentration observed within the first 8 hours of the 24 hour dosing interval.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Median (Full Range); unit: ng/mL
Arm/Group | NuvaRing With ATV/r Plus TDF ≥1 NRTIs
Number analyzed (Participants) | 23
ng/mL
  Cmax day 0 | 4291.0 [769.7 to 9440.0]
  Cmax day 21 | 3583.0 [83.6 to 6578.0]

12. Secondary Outcome: ATV PK Parameter Time to Cmax (Tmax) Determined Based on ATV Levels From Individual Participants Enrolled in Arm C
Description: This evaluates the effect of NuvaRing on the ATV PK parameter Tmax obtained from both sampling periods, before NuvaRing placement (at study day 0) and three weeks later (on study day 21), prior to NuvaRing removal. Tmax defines time to maximum concentration since dose is initiated.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Median (Full Range); unit: hour
Arm/Group | NuvaRing With ATV/r Plus TDF ≥1 NRTIs
Number analyzed (Participants) | 23
hour
  Tmax day 0 | 2.9 [0.9 to 4.0]
  Tmax day 21 | 3.0 [0.0 to 5.0]

13. Secondary Outcome: ATV PK Parameter CLss/F Determined Based on ATV Levels From Individual Participants Enrolled in Arm C
Description: This evaluates the effect of NuvaRing on the ATV PK parameter CLss/F obtained from both sampling periods, before NuvaRing placement (at study day 0) and three weeks later (on study day 21), prior to NuvaRing removal. CLss/f defines apparent oral clearance.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Median (Full Range); unit: L/h
Arm/Group | NuvaRing With ATV/r Plus TDF ≥1 NRTIs
Number analyzed (Participants) | 23
L/h
  CLss/F day 0 | 6.8 [3.3 to 34.1]
  CLss/F day 21 | 8.2 [2.8 to 222.7]

14. Secondary Outcome: Ritonavir (RTV) PK Parameter AUC(0-24h) Calculated Based on Intensive RTV PK Samples Obtained From Individual Participants Enrolled in Arm C
Description: This evaluates the effect of NuvaRing on the PK parameter AUC(0-24h) of RTV before NuvaRing placement (at study day 0) and three weeks later (on study day 21), prior to NuvaRing removal. AUC(0-24h) defines area under the concentration-time curve over the period of 24 hours (pre-dose concentration was used to impute concentration at 24h).
Time Frame: Intensive RTV PK samples at pre-dose, 1, 3, 4, 5, and 8 hours post-dose on study day 0 (before vaginal ring placement) and on study day 21 (3 weeks after vaginal ring placement)
Population: The analysis population is the 23 A5316 participants enrolled in Arm C (NuvaRing with ATV/r arm plus TDF and one or more NRTIs) eligible for the secondary outcome of RTV PK parameters.
Measure: Median (Full Range); unit: h*ng/mL
Arm/Group | NuvaRing With ATV/r Plus TDF and ≥1 NRTIs
Number analyzed (Participants) | 23
h*ng/mL
  AUC0-24h day 0 | 10740.0 [3922.3 to 32632.7]
  AUC0-24h day 21 | 7210.7 [240.0 to 31728.7]

15. Secondary Outcome: RTV PK Parameter Cmin Determined Based on RTV Levels From Individual Participants Enrolled in Arm C
Description: This evaluates the effect of NuvaRing on the PK parameter Cmin of RTV before NuvaRing placement (at study day 0) and three weeks later (on study day 21), prior to NuvaRing removal. Cmin defines minimum concentration observed within the first 8 hours of the 24 hour dosing interval.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Median (Full Range); unit: ng/mL
Arm/Group | NuvaRing With ATV/r Plus TDF and ≥1 NRTIs
Number analyzed (Participants) | 23
ng/mL
  Cmin day 0 | 70.0 [10.0 to 1042.0]
  Cmin day 21 | 51.9 [10.0 to 916.9]

16. Secondary Outcome: RTV PK Parameter Cmax Determined Based on RTV Levels From Individual Participants Enrolled in Arm C
Description: This evaluates the effect of NuvaRing on the PK parameter Cmax of RTV before NuvaRing placement (at study day 0) and three weeks later (on study day 21), prior to NuvaRing removal. Cmax defines maximum concentration observed within the first 8 hours of the 24 hour dosing interval.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Median (Full Range); unit: ng/mL
Arm/Group | NuvaRing With ATV/r Plus TDF and ≥1 NRTIs
Number analyzed (Participants) | 23
ng/mL
  Cmax day 0 | 1437.0 [426.3 to 3078.0]
  Cmax day 21 | 1063.0 [10.0 to 2297.0]

17. Secondary Outcome: RTV PK Parameter Tmax Determined Based on RTV Levels From Individual Participants Enrolled in Arm C
Description: This evaluates the effect of NuvaRing on the PK parameter Tmax of RTV before NuvaRing placement (at study day 0) and three weeks later (on study day 21), prior to NuvaRing removal. Tmax defines time to maximum concentration since dose is initiated.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Median (Full Range); unit: hour
Arm/Group | NuvaRing With ATV/r Plus TDF and ≥1 NRTIs
Number analyzed (Participants) | 23
hour
  Tmax day 0 | 3.0 [0.9 to 5.0]
  Tmax day 21 | 3.0 [0.0 to 5.0]

18. Secondary Outcome: RTV PK Parameter CLss/F Determined Based on RTV Levels From Individual Participants Enrolled in Arm C
Description: This evaluates the effect of NuvaRing on the PK parameter CLss/F of RTV before NuvaRing placement (at study day 0) and three weeks later (on study day 21), prior to NuvaRing removal. CLss/F defines apparent oral clearance.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Median (Full Range); unit: hour
Arm/Group | NuvaRing With ATV/r Plus TDF and ≥1 NRTIs
Number analyzed (Participants) | 23
hour
  CLss/F day 0 | 9.3 [3.1 to 25.5]
  CLss/F day 21 | 13.9 [3.2 to 416.7]

19. Secondary Outcome: Proportion of Participants With Plasma HIV-1 RNA Levels <40 Copies/mL
Description: This evaluates the short-term impact of Nuvaring on virologic suppression in participants who have been administered Nuvaring alone or together with EFV or ATV/r by measuring proportion of participants with plasma HIV-1 RNA levels <40 copies/mL at study day 0 (before vaginal ring placement) and study day 21 (three weeks after vaginal ring placement). An FDA-approved HIV-1 RNA assay was required.
Time Frame: Study day 0 and study day 21
Population: All participants in whom NuvaRing was inserted and with HIV-1 RNA data available.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | NuvaRing and no ART | NuvaRing With EFV Plus ≥2 NRTIs | NuvaRing With ATV/r Plus TDF and ≥1 NRTIs
Number analyzed (Participants) | 27 | 28 | 28
proportion of participants
  Proportion with HIV-1 RNA <40 copies/mL at day 0: number analyzed (Participants) | 23 | 27 | 28
  Proportion with HIV-1 RNA <40 copies/mL at day 0 | 0.22 [0.07 to 0.44] | 0.93 [0.76 to 0.99] | 0.89 [0.72 to 0.98]
  Proportion with HIV-1 RNA <40 copies/mL at day 21: number analyzed (Participants) | 24 | 26 | 27
  Proportion with HIV-1 RNA <40 copies/mL at day 21 | 0.17 [0.05 to 0.37] | 0.85 [0.65 to 0.96] | 0.85 [0.66 to 0.96]

20. Secondary Outcome: Percentage of Participants With Signs and Symptoms of Grade 2 or Higher Deemed Possibly, Probably or Definitely Related to Study Treatment
Description: This evaluates toxicity and safety of NuvaRing alone, NuvaRing with EFV, and NuvaRing with ATV/r. Signs/symptoms were graded using the DAIDS AE Grading Table was used. Participants with sign(s)/symptom(s) of grade 2 (moderate), 3 (severe), 4 (potentially life-threatening) or 5 (death) are included in the percentage. Relationship to study treatment was determined by the study co-chairs and DAIDS clinical representative.
Time Frame: From day 0 to day 28
Population: All participants in whom NuvaRing was inserted
Measure: Number; unit: Percent of Participants
Arm/Group | NuvaRing and no ART | NuvaRing With EFV Plus ≥2 NRTIs | NuvaRing With ATV/r Plus TDF and ≥1 NRTIs
Number analyzed (Participants) | 27 | 28 | 28
Percent of Participants | 7.4 | 3.6 | 3.6

21. Secondary Outcome: Proportion of Participants With Progesterone Levels Greater Than 5 ng/mL.
Description: This evaluates alterations in progesterone levels due to the potential PK interaction between NuvaRing and the ARVs EFV and ATV/r by examining progesterone levels at study days 0 (before vaginal ring placement), 7, 14, and 21 (before vaginal ring removal), and study day 28, without regard to menstrual cycle status at study entry.
Time Frame: Study days 0, 7, 14, 21 and 28
Population: All participants included in the primary analyses who had progesterone data available. One participant on the EFV arm is excluded at day 14 visit because NuvaRing was out of the body for >3 hours leading up to the visit.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | NuvaRing and no ART | NuvaRing With EFV Plus ≥2 NRTIs | NuvaRing With ATV/r Plus TDF and ≥1 NRTIs
Number analyzed (Participants) | 25 | 25 | 24
proportion of participants
  Proportion with progesterone >5 at day 0 | 0.08 [0.01 to 0.26] | 0.04 [0.00 to 0.20] | 0.25 [0.10 to 0.47]
  Proportion with progesterone >5 at day 7: number analyzed (Participants) | 24 | 25 | 24
  Proportion with progesterone >5 at day 7 | 0.08 [0.01 to 0.27] | 0.24 [0.09 to 0.45] | 0.08 [0.01 to 0.27]
  Proportion with progesterone >5 at day 14: number analyzed (Participants) | 24 | 24 | 24
  Proportion with progesterone >5 at day 14 | 0.00 [0.00 to 0.14] | 0.04 [0.00 to 0.21] | 0.00 [0.00 to 0.14]
  Proportion with progesterone >5 at day 21 | 0.00 [0.00 to 0.14] | 0.00 [0.00 to 0.14] | 0.00 [0.00 to 0.14]
  Proportion with progesterone >5 at day 28: number analyzed (Participants) | 24 | 24 | 24
  Proportion with progesterone >5 at day 28 | 0.00 [0.00 to 0.14] | 0.00 [0.00 to 0.14] | 0.00 [0.00 to 0.14]

ADVERSE EVENTS:
Time Frame: From Day 0 to Day 28.
Description: Protocol required reporting: diagnoses (identified by ACTG criteria for clinical events and other diseases); signs/symptoms of grade ≥3; selected signs/symptoms of grade ≤2 (gynecological and/or deemed related to the NuvaRing or study procedures); hematology, LFTs and chemistry findings of grade ≥2. The DAIDS AE Grading Table and Version 2.0 of the DAIDS EAE Manual were used. One participant on ATV/r arm was excluded from AE analyses because insertion of NuvaRing could not be confirmed.
Arm/Group | NuvaRing and no ART | NuvaRing With EFV Plus ≥2 NRTIs | NuvaRing With ATV/r Plus TDF and ≥1 NRTIs
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 10/27 | 20/28 | 18/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NuvaRing and no ART (N=27) | NuvaRing With EFV Plus ≥2 NRTIs (N=28) | NuvaRing With ATV/r Plus TDF and ≥1 NRTIs (N=28)
Bacterial vaginosis (Infections and infestations) | 1 | 3 | 1
Vulvovaginal candidiasis (Infections and infestations) | 1 | 2 | 0
Blood bicarbonate decreased (Investigations) | 0 | 2 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 3
Blood glucose increased (Investigations) | 2 | 0 | 1
Blood sodium decreased (Investigations) | 3 | 3 | 2
Menstruation normal (Investigations) | 1 | 5 | 8
Libido decreased (Psychiatric disorders) | 0 | 0 | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 1 | 2
Metrorrhagia (Reproductive system and breast disorders) | 1 | 2 | 1
Vaginal discharge (Reproductive system and breast disorders) | 4 | 8 | 4
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 4 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 2 | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.